CLINICAL TRIAL: NCT00541879
Title: Type 2 Diabetes Knowledge: Obesity and Diabetes Prevention Through Science Enrichment
Brief Title: Obesity and Diabetes Prevention Through Science Enrichment
Acronym: DKENERGY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH); Poudre School District, Fort Collins, CO (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H 04-257 RR25 RR 020469; R 25 RR 020469; R 25 RR 015646
Record Dates: First submitted 2007-10-09; First posted 2007-10-10 (Estimated); Last update posted 2014-11-07 (Estimated); Status verified 2014-11

CONDITIONS: Type 2 Diabetes; Obesity
Keywords: Childhood; Prevention; Energy balance; Glucose regulation; Healthy lifestyle; Healthy eating; Active living
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- I (Experimental): Elementary school children -grades 2-6 participating in Program ENERGY
  Interventions: Behavioral: Program ENERGY
- II (Sham Comparator): Elementary school children in grades 2-6 matched to the intervention classes not receiving any intervention
  Interventions: Other: comparison

INTERVENTIONS:
Behavioral: Program ENERGY — Weekly or biweekly classroom and gym based science enrichment focused on how the body works including blood glucose regulation, healthy eating and physical activity, diabetes abd how it can be prevented
  Arms: I
Other: comparison
  Arms: II

SUMMARY:
Type 2 diabetes and obesity in children continue to increase at alarming rates with devastating results. However, both these metabolic diseases are largely preventable through adoption of a healthy lifestyle, an understanding of what happens to food in the body, energy balance and some simple aspects of glucose regulation. Can elementary school children be taught the knowledge and skills necessary to prevent type 2 diabetes and obesity? Children need to learn this essential knowledge and practice these important health behavior skills. Elementary school may be an ideal place to master this subject that is a direct and logical extension of current health curricula including nutrition and physical activity blended with science and math.

DETAILED DESCRIPTION:
Biomedical scientists lead a classroom series of interactive, inquiry-based science and health explorations directed at type 2 diabetes, obesity and their prevention in three elementary schools serving children at high risk for type 2 diabetes. Diabetes knowledge was measured in children and parents at the beginning, end and 9 months after the end of the intervention using validated questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Elementary school child in selected intervention or comparison classes/schools

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2909 (Actual)
Dates: Start 2001-08; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Diabetes knowledge and prevention behaviors in elementary school children | one-three school year(s)

SECONDARY OUTCOMES:
Parental diabetes knowledge, self-reported physical activity | one -three school year(s)

CONTACTS AND LOCATIONS:
Overall Officials: L. Arthur Campfield, PhD, Principal Investigator — Colorado State University
Locations (1):
- Putnam, Tavelli, Bennett and Dunn Elementary Schools, Fort Collins, Colorado, United States

REFERENCES:
- See also: Program ENERGY website — http://www.ProgramENERGY.org